CLINICAL TRIAL: NCT01324427
Title: Pilot Trial of Telemedicine Evaluation for Stem Cell Transplant Patients
Brief Title: Telemedicine Evaluation for Stem Cell Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-022
Record Dates: First submitted 2011-03-24; First posted 2011-03-29 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Stem Cell Transplant Patients
Keywords: Telemedicine; Virtual Medical Visit; Quality of Life; 11-022

ARMS (1):
- virtual medical visit (Experimental): This is a pilot trial involving a maximum of 84 patients undergoing either allogeneic or autologous stem cell transplant aimed at determining the feasibility and acceptance of a "virtual medical visit" by patients and health care personnel. During this pilot trial we expect to perform 84 "virtual medical visits" using telemedicine.
  Interventions: Behavioral: virtual medical visit

INTERVENTIONS:
Behavioral: virtual medical visit — At the pre-set time, the "Mobile Telehealth Cart" will be set up in the exam room or the clinic office, and a connection with the doctor will be made through their computer. The telemedicine visit will be conducted at the same time as the regular clinic visit. During the visit, the nurse will evaluate the physical symptoms, vital signs, past medical history, present medical history, and any side effects from the autologous or allogeneic transplant. The nurse will place a digital stethoscope on the chest to listen to the heart and lungs. The "virtual medical visit" will take about 25 minutes. At the end of the "Virtual Medical Visit," the patient will evaluate the event using a survey to assess the acceptance of the virtual visit. The surveys will be written and should take around 15 minutes to complete. The answers provided will be shared with the MD and nurses after the patient has completed all their "virtual medical visits."

SUMMARY:
Telemedicine is a new area of health care where medical information is transferred through audiovisual media, such as a computer or a video camera, for the purpose of remote doctor's visits or examinations. This new area of health care is important to test because it can potentially provide real-time interactions between the patient and their health care team, including phone conversations, online communication, and/or home visits. Many activities such as a history review or physical examination can be conducted virtually as compared to the traditional face-to face visits.

The purpose of this study is to determine patient and health care team acceptance of a "virtual medical visit" as a substitute for a "face to face" visit for patients either preparing to receive a stem cell transplant or previously received a stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent or are planning to undergo a hematopoietic progenitor cell transplantation for any disease.
* Participants must be able to read and understand English*
* Age over 18 years of age since this pilot trial is only being performed in the Adult BMT Service Non-English speaking patients have been excluded in this pilot study because we do not have the support for translation services at this time. Additionally, the telemedicine instruments being used are not yet validated across all languages.

Potential patients will be identified according to their medical condition, type and complexity of stem cell transplant procedure performed, and distance from MSKCC.

The patients should:

1. minimal comorbidities,
2. be less than 75 years of age. These characteristics have been associated with good understanding and acceptance of telemedicine in other pilot trials. These characteristics will be assessed by the clinician.

Please note: Patients on other therapeutic protocols will be eligible for this protocol as well.

Exclusion Criteria:

* Medically unstable patient as deemed by the treating team.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2011-03; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Determine patient & physician acceptance of a "virtual medical visit" as a substitute for a "face to face" in pts in different settings. This is assessed by analyzing answers to questions 7 & 8 of the Patient Satisfaction Survey. [Question #7: I would | 2 years
  Question #8: Overall, I was very satisfied with today's telemedicine session.]Physician acceptance will be analyzed looking at the answers to question 19 of the Physician/Nurse survey in which the physician or nurse investigator relates the quality of the telemedicine visit. [Question #19: How would you rate the quality of the Telehealth visit to assess the patient compared to an in-person office visit?]

SECONDARY OUTCOMES:
Confirm that current telemedicine technology a comprehensive stem cell transplant clinical evaluation can be performed. | 2 years
  Questions 1-12 of the healthcare provider survey will assess the quality of the information &assessment collected through the "virtual medical visit".
Evaluate the feasibility of telemedicine facilitated "handoffs" between the inpatient and the outpatient service at the time of discharge from the inpatient service and at the time of discharge from the transplant center are feasible and useful. | 2 years
  The instrument used to analyze the feasibility and utility of the handoff instrument is Provider Satisfaction Survey with Handoff Instrument Survey for Feedback on Handoff Instrument. We will collate these responses to determine whether the handoff instrument was found to be useful and what elements should be modified, removed or added.
Describe the logistic characteristics of a "virtual medical visit" performed using telemedicine such as visit times, connection quality, and quality of the clinical information obtained. | 2 years
  The time from the first attempt to connect until the time to disconnect will be captured for all encounters as well as the time from the beginning to end of the "virtual medical visit". We expect that the "virtual medical visit" should take on average 20 minutes from attempt to connect to disconnect.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Giralt, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm